CLINICAL TRIAL: NCT01820585
Title: Efficacy and Safety of Eslicarbazepine Acetate as Therapy in Subjects With Fibromyalgia: a Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Therapy in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-2093-210
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-06

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; Eslicarbazepine acetate (BIA 2-093); ESL
MeSH Terms: conditions — Fibromyalgia | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Tablets
  Interventions: Drug: Placebo
- ESL 400 mg (Active Comparator): Eslicarbazepine acetate (BIA 2-093) tablets
  Interventions: Drug: ESL 400 mg
- ESL 800 mg (Active Comparator): Eslicarbazepine acetate (BIA 2-093) tablets
  Interventions: Drug: ESL 800 mg
- ESL 1200 mg (Active Comparator): Eslicarbazepine acetate (BIA 2-093) tablets
  Interventions: Drug: ESL 1200 mg

INTERVENTIONS:
Drug: Placebo — Tablets
  Other Names: Sugar pills
  Arms: Placebo
Drug: ESL 400 mg — tablets
  Other Names: Eslicarbazepine acetate (BIA 2-093)
  Arms: ESL 400 mg
Drug: ESL 800 mg — tablets
  Other Names: Eslicarbazepine acetate (BIA 2-093)
  Arms: ESL 800 mg
Drug: ESL 1200 mg — tablets
  Other Names: Eslicarbazepine acetate (BIA 2-093)
  Arms: ESL 1200 mg

SUMMARY:
This was a double-blind, randomised, placebo-controlled, parallel-group, multicentre, multinational, Phase II study in 528 subjects with pain due to Fibromyalgia syndrome(FMS). Subjects were randomised in a 1:1:1:1 ratio to receive placebo, Eslicarbazepine acetate (ESL) 400 mg once daily (QD), ESL 800 mg QD or ESL 1200 mg QD. The study was carried out as follows.

DETAILED DESCRIPTION:
This was a double-blind, randomised, placebo-controlled, parallel-group, multicentre, multinational, Phase II study in 528 subjects with pain due to FMS. Subjects were randomised in a 1:1:1:1 ratio to receive placebo, ESL 400 mg once daily (QD), ESL 800 mg QD or ESL 1200 mg QD. The study was carried out as follows:

Screening Visit (Visit [V] 1): After completing screening procedures at V1, eligible subjects began the 2 week Baseline Period.

Baseline Period (2 weeks): Subjects discontinued taking prohibited medications on V1 (beginning of washout period). Subjects were tapered off of discontinued medications. Washout was completed by Day -7 (7 days before V2). Subjects refrained from taking any pain medications and other prohibited medications (except rescue medication) throughout the study. During the Baseline Period, subjects used the subject diary to complete the diary pain assessment on a 0-10 numeric pain rating scale (NPRS) and to record information on rescue medication daily on awakening.

Titration Period (1 week): Upon completing the Baseline Period, subjects returned to the study centre for V2 (Randomisation Visit, Day 1). At V2, subjects, who had completed at least 4 subject diary pain assessments satisfactorily within the past 7 days, had an average pain score that was ≥4 and ≤9 and continued to meet all study entry criteria, were randomly assigned to 1 of the 4 treatment groups. During the 1-week Titration Period, subjects randomised to the ESL 400 mg QD and the ESL 800 mg QD treatment groups received ESL 400 mg QD; and subjects randomised to the ESL 1200 mg QD treatment group received ESL 600 mg QD; subjects assigned to placebo treatment received placebo QD.

Maintenance Period (12 weeks): Starting at V3, subjects assigned to treatment with ESL received their full dosage regimens QD; subjects assigned to placebo treatment received placebo QD. During the Maintenance Period, subjects had visits every 4 weeks.

Follow-up Period (2 weeks): Approximately 2 weeks after taking the last dose of study medication, subjects returned to the study centre for the Follow-up Visit and underwent the end-of-study evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Subject was male or female, 18 years of age or older (according to Amendment #1 for Czech Republic [24 MARCH 2009]: 18 to 65 years of age).
* Subject was able and willing to provide written informed consent to participate in the study after having the opportunity to review the Subject Information Sheet and Informed Consent Form.
* Subject met the American College of Rheumatology (ACR) 1990 diagnostic criteria for FMS (widespread pain for at least 3 months and pain in at least 11 of 18 tender points) (according to Amendment #1 for Czech Republic [24 MARCH 2009]: and the subject's current FMS treatment was either inefficacious or had intolerable side effects).
* Subject was willing and able to understand and comply with all study requirements, in the judgment of the investigator.
* Subject had negative results on the urine test for drugs of abuse at V1 (Screening Visit), except for medications/drugs reported by the subject at the Screening Visit.
* Subject use of allowable non-pharmacological therapies was stable for at least 4 weeks prior to V1 (Screening Visit) and would be maintained at the stable regimen throughout the study.
* Female subject was surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or at least 2 years post-menopausal or, if of childbearing potential, she was sexually abstinent or agreed to use a medically acceptable non-hormonal method of contraception
* Addendum according to Amendment #1 for Czech Republic [24 MARCH 2009]: Hormonal contraceptives were not acceptable as a contraceptive method in this study. However, their intake was not forbidden throughout the study.
* Addendum according to Amendment #1 for Spain [19 JANUARY 2009] and for United Kingdom [24 MARCH 2009]: Male subject was sexually abstinent or agreed to use reliable contraceptive methods (i.e. double-barrier method: 1 male barrier [male condom] plus 1 female barrier method [female condom, spermicide or intrauterine device]. This was mandatory even for sexually active men who had been sterilised.
* Subject had a negative urine test for drugs of abuse.
* The subject had completed at least 4 subject diary pain assessments satisfactorily within the past 7 days prior to V2 and the average pain score was ≥4 and ≤9.

Exclusion Criteria:

* Subject had a known hypersensitivity to ESL or to other carboxamide derivatives (e.g. oxcarbazepine, carbamazepine) or to any of the excipients.
* Subject had a history of or current active malignancy except for the following: basal cell carcinoma which had been treated; and malignancies that were successfully treated and had no recurrence within 5 years before V1 (Screening Visit).
* Subject had a severe hepatic, renal, respiratory, hematologic or immunologic illness, unstable cardiovascular disease or any other medical or psychiatric condition that, in the judgment of the investigator, made the subject inappropriate for entry into this study.
* Subject had a second or third-degree atrioventricular blockade not corrected with a pacemaker or any other clinically significant abnormality in the 12-lead ECG as determined by the investigator.
* Subject had a history of illicit drug or alcohol abuse within 2 years before V1 (Screening Visit).
* Subject had received an investigational drug (or a medical device) within 3 months of Screening or was currently participating in another study of an investigational drug (or a medical device).
* Subject was pregnant or nursing.
* Subject was an employee of the investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that investigator or study centre or was a family member of the employees or the investigator.
* Subject had any of the following: an inflammatory muscle or rheumatologic disease other than FMS; multiple sclerosis; active infections; untreated endocrine disorders; uncontrolled hypo- or hyper-thyroidism of any type.
* Subjects whose pain was not due primarily to FMS.
* Subject underwent tender point injection within 30 days before V1 (Screening Visit) and/or subject was unwilling to refrain from tender point injection throughout the study.
* Subject had a white blood cell (WBC) count <2.5 × 109/L, neutrophil count <1.5 × 109/L, Na+ <125 mmol/L or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 × the upper limit of normal at V1 (Screening Visit) or any other clinically relevant laboratory abnormality that, in the investigator's opinion, could compromise the subject's safety.
* Subject had abnormal values for antinuclear antibody (ANA >1/160) or rheumatoid factor (RF >15 IU/mL) at V1 (Screening Visit). After approval of the global amendment in respective countries, the limit for ANA was changed to ≥1/160.
* Subject had abnormal Westergren erythrocyte sedimentation rate (ESR) at V1 (Screening Visit) (ESR >40 mm/h).
* Subject had creatinine clearance (CLCr) lower than 60 mL/min at Screening.
* Subject had a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≥35 or a score of 4 to 6 on question 10 of the MADRS at V1 (Screening Visit).
* Subject used prohibited concomitant medications during the 2-week Baseline Period or used fluoxetine during the 30 days before V1 (Screening Visit).
* Subject used opiates every day for the 30 days before V1 (Screening Visit) for the control of pain related to FMS.
* Exclusion criterion at V2:
* Subject had a MADRS total score ≥35 or a score of 4 to 6 on question 10 of the MADRS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Cª, S.A.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened in 84 centres in 16 European countries (Austria, Bulgaria, Czech Republic, France, Germany, Hungary, Italy, Netherlands, Poland, Portugal, Romania, Serbia, Slovakia, Spain, Ukraine and United Kingdom).
  Study initiation date: 21 Apr 2009 Study completion date: 03 Sep 2010;
Pre-assignment Details: After completing procedures at V1, subjects returned to the study centre for V2. At V2, subjects, who had completed at least 4 subject diary pain assessments satisfactorily within the past 7 days, had an average pain score that was ≥4 and ≤9 and continued to meet all study entry criteria, were randomly assigned to 1 of the 4 treatment groups.
Groups:
- Placebo: Placebo tablets matching the 400-mg and 600-mg tablets were administered Once daily (QD) by oral route.
- ESL 400 mg: Eslicarbazepine acetate (ESL) 400 mg : ESL was supplied in 400-mg tablets and was administered QD by oral route.
- ESL 800 mg: ESL 800 mg : ESL was supplied in 400-mg tablets and was administered QD by oral route
- ESL 1200 mg: ESL was supplied in 400-mg and 600-mg tablets and was administered QD by oral route.
Period: Overall Study
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg
Started | 131 | 130 | 135 | 132
Randomized and Treated | 131 | 130 | 135 | 132
Full Analysis Set | 131 | 130 | 135 | 129
Completed Titration Period | 128 | 125 | 131 | 126
Entered Maintenance Period | 128 | 124 | 131 | 123
Completed Maintenance Period | 105 | 98 | 101 | 84
Completed | 104 | 98 | 101 | 83
Not Completed | 27 | 32 | 34 | 49
Not completed — Adverse Event | 9 | 13 | 23 | 34
Not completed — Lack of Efficacy | 9 | 7 | 5 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 3 | 8
Not completed — Lost to Follow-up | 3 | 3 | 0 | 3
Not completed — Protocol Violation | 3 | 1 | 1 | 1
Not completed — Subject non-compliance | 0 | 0 | 1 | 2
Not completed — at sponsor request | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Tablets
  Placebo : Tablets
- ESL 400 mg: Eslicarbazepine acetate (BIA 2-093) tablets
  ESL 400 mg : Eslicarbazepine acetate (BIA 2-093) tablets
- ESL 800 mg: Eslicarbazepine acetate (BIA 2-093) tablets
  ESL 800 mg : Eslicarbazepine acetate (BIA 2-093) tablets
- ESL 1200 mg: Eslicarbazepine acetate (BIA 2-093) tablets
  ESL 1200 mg : Eslicarbazepine acetate (BIA 2-093) tablets
- Total: Total of all reporting groups
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg | Total
Number analyzed (Participants) | 131 | 130 | 135 | 132 | 528
Age, Customized [Number; unit: participants]
  <=65 Years | 126 | 126 | 132 | 127 | 511
  >65 years | 5 | 4 | 3 | 5 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 114 | 127 | 122 | 487
  Male | 7 | 16 | 8 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Endpoint in Mean Pain
Description: The primary efficacy variable was the absolute change from baseline to endpoint in mean pain. Pain intensity was assessed on an 11-point (0-10) Numeric pain rating scale (NPRS), where 0 = no pain and 10 = worst possible pain and was recorded in a subject's diary. The subject was instructed to complete the assessment daily on awakening.Primary analyses were conducted on the full analysis set (FAS) which consisted of all randomised subjects who received at least 1 dose of study medication and with at least 1 post-randomisation rating of 24-h-average pain. The primary efficacy variable was the absolute change from baseline to endpoint in mean pain recorded in a subject's diary upon awakening each morning. An ANCOVA on the FAS revealed no statistically significant differences between the 3 ESL groups and the placebo group after 13 weeks of treatment.
Time Frame: Baseline and 13 Weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg
Number analyzed (Participants) | 130 | 130 | 135 | 129
units on a scale | -1.0 (0.1735) | -0.8 (0.1731) | -1.2 (0.1704) | -0.8 (0.1734)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were evaluated throughout the study that consisted of a 2-week Baseline Period, a 1-week Titration Period (active treatment or placebo) and a 12- week Maintenance Period (active treatment or placebo).
Description: Safety was evaluated based on adverse events (AEs)
Arm/Group | Placebo | ESL 400 mg | ESL 800 mg | ESL 1200 mg
Serious Adverse Events (participants affected / at risk) | 3/131 | 5/130 | 6/135 | 1/132
Other Adverse Events (participants affected / at risk) | 75/131 | 86/130 | 92/135 | 93/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=131) | ESL 400 mg (N=130) | ESL 800 mg (N=135) | ESL 1200 mg (N=132)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=131) | ESL 400 mg (N=130) | ESL 800 mg (N=135) | ESL 1200 mg (N=132)
Headache (Nervous system disorders) | 16 (16) | 18 (18) | 19 (19) | 25 (25)
Nausea (Gastrointestinal disorders) | 10 (10) | 10 (10) | 17 (17) | 21 (21)
Dizziness (Nervous system disorders) | 6 (6) | 7 (7) | 7 (7) | 15 (15)
Fatigue (General disorders) | 5 (5) | 5 (5) | 7 (7) | 11 (11)
Gamma-glutamyl transferase increased (Investigations) | 0 (0) | 6 (6) | 8 (8) | 10 (10)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 5 (5) | 9 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (4) | 9 (9)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 14 (14) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 8 (8) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 6 (6) | 5 (5) | 8 (8)
Somnolence (Nervous system disorders) | 4 (4) | 3 (3) | 3 (3) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (6) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 4 (4) | 4 (4)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 3 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 3 (3) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (4)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (4) | 3 (3) | 1 (1)
Pain (General disorders) | 3 (3) | 2 (2) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other